CLINICAL TRIAL: NCT01948765
Title: Xenon as an Adjuvant to Propofol Anaesthesia in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery:a Randomised Controlled Trial
Brief Title: Xenon as an Adjuvant to Propofol Anaesthesia in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof Dr Steffen Rex, PhD, MD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR022013
Record Dates: First submitted 2013-08-08; First posted 2013-09-24 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease; Anesthesia
Keywords: xenon anesthesia; Off-pump coronary artery bypass graft surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Xenon; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon and propofol (Active Comparator)
  Interventions: Drug: Xenon and propofol
- propofol (Placebo Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Xenon and propofol — xenon 30% in oxygen as an adjuvant to propofol target controlled infusion (target of 0.5-1.5µg/ml)
  Arms: Xenon and propofol
Drug: propofol — propofol target controlled infusion (target 1.5-2.5µg/ml)
  Arms: propofol

SUMMARY:
The investigators hypothesize that the application of 30% xenon as an adjuvant to general anesthesia with a target-controlled infusion of propofol is superior to general anesthesia with propofol alone with respect to hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease scheduled for elective OPCAB-surgery
* patients willing and able to complete the requirements of this study
* Ejection fraction >30%

Exclusion Criteria:

* Lack of informed consent
* age < 18 years
* COPD GOLD >II
* Renal dysfunction defined as serum-creatinine >1.5mg/dl
* acute coronary syndrome during the last 24 hours; haemodynamic instability, requirement of inotropic support
* single vessel grafting
* disabling neuropsychiatric disorders (severe dementia, Alzheimer's disease, schizophrenia, depression, low preoperative cognitive state (MMSE at baseline <25), history of stroke with residuals, increased intracranial pressure
* Hypersensitivity to the study medication
* Presumed uncooperativeness or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
intraoperative haemodynamic stability | intra-operative
  Haemodynamic stability as assessed by the individual intraoperative noradrenaline consumption

SECONDARY OUTCOMES:
MACCE (major adverse cardiac and cerebral events) | up to six months postoperative
  Death from any cause, perioperative life-threatening cardiac arrhythmias, perioperative myocardial infarction, requirement of surgical revisions at the coronary vessels, postoperative coronary angioplasty and stroke
cerebrovascular accident not included in MACCE | up to six months postoperative
  cerebrovascular accident not included in MACCE (TIA, reversible ischaemic neurologic deficit)
postoperative renal function | up to five days postoperative
  postoperative renal function as assessed by serum creatinine and BUN levels)
requirement for blood(product) transfusion | up to five days postoperative
  requirement for blood(product) transfusion
length of stay | participants will be followed for the duration of hospital stay, an expected average of 10 days.
  requirement for blood(product) transfusion
severity of postoperative critical illness | up to five days postoperative
  Severity of postoperative critical illness as indicated by the new simplified acute physiology score (SAPS II), SOFA and APACHE-II score
incidence and duration of postoperative delirium | participants will be followed for the duration of hospital stay, an expectged average of 10 days
  incidence and duration of postoperative delirium assessed with the Confusion Assessment Method (CAM-ICU), to be assessed in combination with the Mini Mental State Examination
incidence of further AE, SAE and SUSAR | participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Al Tmimi L, Devroe S, Dewinter G, Van de Velde M, Poortmans G, Meyns B, Meuris B, Coburn M, Rex S. Xenon as an Adjuvant to Propofol Anesthesia in Patients Undergoing Off-Pump Coronary Artery Bypass Graft Surgery: A Pragmatic Randomized Controlled Clinical Trial. Anesth Analg. 2017 Oct;125(4):1118-1128. doi: 10.1213/ANE.0000000000002179. PMID 28598913